CLINICAL TRIAL: NCT01101113
Title: Phase 4 Study of Cinacalcet Efficacy in Combination With Vitamin D for the Treatment of Secondary Hyperparathyroidism in Peritoneal Dialysis Patients
Brief Title: Cinacalcet stUdy for Peritoneal Dialysis Patients In Double Arm on the Lowing Effect OF iPTH Level
Acronym: CUPID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Jeil-Kirin Pharmaceutical Inc. (Industry)
Responsible Party: Principal Investigator, Kook-Hwan Oh, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINA-Kor-01
Record Dates: First submitted 2010-04-04; First posted 2010-04-09 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Secondary Hyperparathyroidism
Keywords: peritoneal dialysis
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cinacalcet (Experimental): stepwise dose of cinacalcet + regular medical medication including vit D
  Interventions: Drug: cinacalcet
- Control (Active Comparator): conventional treatment for secondary HPT including vit D and phosphate binder
  Interventions: Drug: control

INTERVENTIONS:
Drug: cinacalcet — cinacalcet 25mg qd or 50 mg qd
  Arms: Cinacalcet
Drug: control — vit D + P binder
  Arms: Control

SUMMARY:
This study is designed in order to investigate the effect of cinacalcet in combination with routine conventional medical management for treatment of secondary hyperparathyroidism (SHPT) and Ca, P control. This study will compare the efficacy of a cinacalcet-based regimen with unrestricted conventional care (vitamin D and phosphate binders) for achieving the stringent National Kidney Foundation Kidney Disease Outcomes Quality Initiative (KDOQI) targets for dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Peritoneal dialysis patients with secondary HPT(iPTH > 300 pg/mL)
* > 18 yr of age, < 70
* had receive PD for > 3 mo,
* intact PTH level > 300 pg/ml and <1000 pg/ml
* albumin corrected Ca level >= 9.0 mg/dL

Exclusion Criteria:

* pregnant or breast-feeding,
* had undergone parathyroidectomy within previous 3 mo,
* are involved in other clinical trial within 30 d
* had received cinacalcet therapy previously.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
> 30% reduction from baseline of intact parathyroid hormone (iPTH) | 20 weeks

SECONDARY OUTCOMES:
Achievement of treatment goal of intact parathyroid hormone (iPTH) (150~300 pg/ml) | 20 weeks
Achievement of targets for mean Ca x P (<55 mg2/dL2), Ca (<9.5 mg/dL), P (<5.5 mg/dL) | 20 weeks
Achieving targets for intact PTH (150-300 pg/ml) and calcium-phosphorus product (Ca x P) (<55 mg2/dl2) simultaneously | 20 weeks
Vascular calcification score | 20 weeks
  Abdominal aortic calcification score (AAC, 0-24) will be measured at baseline and at 20 weeks according to Kauppila et al (Atherosclerosis 2004)
Normalization of serum alkaline phosphatase | 20 weeks
  Serum alkaline phosphatase measured at baseline and 20 weeks
Serum FGF-23 | baseline and 20th week
  Elevated serum levels of fibroblast growth factor-23 (FGF23) is associated with adverse outcomes in dialyzed patients. Therefore, we added analysis of change in FGF23 levels between two treatments to explore the cinacalcet effect in lowering FGF23.

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Seoul National University Hospital, Seoul, Korea
  - Kyungpook National University, Daegu
  - Gil Hospital, Incheon
  - Hallym University Sacred Hospital, Pyungchon
  - Seoul National University Bundang Hospital, Seongnam
  - Eulji University, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Kim HJ, Kim H, Shin N, Na KY, Kim YL, Kim D, Chang JH, Song YR, Hwang YH, Kim YS, Ahn C, Lee J, Oh KH; Representing the Cinacalcet stUdy for Peritoneal Dialysis Patients In Double Arm on the Lowing Effect Of iPTH Level (CUPID) Study Group. Cinacalcet lowering of serum fibroblast growth factor-23 concentration may be independent from serum Ca, P, PTH and dose of active vitamin D in peritoneal dialysis patients: a randomized controlled study. BMC Nephrol. 2013 May 25;14:112. doi: 10.1186/1471-2369-14-112. PMID 23705925